CLINICAL TRIAL: NCT06953674
Title: Saline vs. Balanced Crystalloid in Traumatic Brain Injury
Brief Title: Saline Versus Balanced Crystalloid in Traumatic Brain Injury
Acronym: FLUID-TBI
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: Kentucky Spinal Cord and Head Injury Research Board (Unknown)
Responsible Party: Principal Investigator, Akshitkumar MIstry, Assistant Professor Term, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24.0224
Record Dates: First submitted 2025-04-09; First posted 2025-05-01 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Traumatic Brain Injury (TBI) Patients
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Normal Saline (Experimental): normal saline (0.9% sodium chloride) administered intravenously
  Interventions: Drug: Normal Saline (0.9% NaCl)
- Isotonic Crystalloid (Active Comparator): balanced crystalloid intravenous fluid therapy
  Interventions: Drug: balanced crystalloid

INTERVENTIONS:
Drug: Normal Saline (0.9% NaCl) — For the primary purpose of fluid therapy or resuscitation in the emergency room and during hospitalization. The interventions will be administered intravenously whenever isotonic intravenous fluid administration is ordered by the treating provider for fluid resuscitation and/or maintenance in the emergency room and during inpatient hospitalization. Assignment to the intervention arm will be adhered to from enrollment to discharge. The total volume, rate, initiation, cessation, and co-interventions will be left to the discretion of the treating provider. Adherence will be ensured by dual interventions at the level of pharmacy IV fluid supply and physician order. The fluids will be physically administered according to the standard intravenous procedures and those outlined in the manufacturer's instructions.
  Arms: Normal Saline
Drug: balanced crystalloid — For the primary purpose of fluid therapy or resuscitation in the emergency room and during hospitalization. The interventions will be administered intravenously whenever isotonic intravenous fluid administration is ordered by the treating provider for fluid resuscitation and/or maintenance in the emergency room and during inpatient hospitalization. Assignment to the intervention arm will be adhered to from enrollment to discharge. The total volume, rate, initiation, cessation, and co-interventions will be left to the discretion of the treating provider. Adherence will be ensured by dual interventions at the level of pharmacy IV fluid supply and physician order. The fluids will be physically administered according to the standard intravenous procedures and those outlined in the manufacturer's instructions.
  Arms: Isotonic Crystalloid

SUMMARY:
The goal of this clinical trial is to determine which crystalloid (saline or balanced) should be used in the critical management of Traumatic Brain Injury (TBI) in moderate or severe TBI patients. This trial will determine whether the use of saline or balanced crystalloids is associated with improved outcomes in TBI patients.

Participants will

1. be given fluids through the veins, either saline or balanced fluid will be given.
2. From the first day to the day 14 of the hospitalization (or discharge, whichever comes first), vital signs, laboratory values, treatments given, and other medical data will be collected from the medical record.
3. Six months later, your final disability, if any, will be assessed during your follow-up with a doctor. It involves answering a short survey that will take about 5 minutes or less.

ELIGIBILITY:
Inclusion Criteria:

* Trauma patients presenting to the Emergency Room for initial care
* Glasgow Coma Scale ≤ 12
* Head CT with skull fracture(s) and/or hemorrhage(s) (>1cm in any single dimension) with a reported mechanism of trauma

Exclusion Criteria:

* Severe visceral trauma dictating mortality (visceral injury severity score > brain injury severity score)
* Non-survivable brain injury based on the treating physician's judgment
* Emergent visceral operative intervention before complete trauma assessment
* Concern for ruptured intracranial vascular malformation
* Patients who are transferred from another facility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Neurological Outcomes | 6 months post injury
  Glasgow Outcome Scale-Extended (GOSE) 8-point scale. Glasgow Outcome Scale has been widely accepted as the standard assessment scale of global outcomes after severe brain injury because it captures well how the injury affects functioning in major areas of life. Using the manual for the GOSE interview, we will conduct our primary efficacy assessment at 6 months after ICU admission in person or over the phone. Outcomes on the GOSE scale do not change past the 6-month mark in moderate and severe TBI patients.
  The 8-point ordinal GOSE scale for the primary efficacy assessment will be dichotomized into favorable (GOSE score 4-8) and unfavorable (GOSE 1-3) outcomes. The primary analysis model will be a logistic regression model where the outcome of interest is the dichotomized GOS-E evaluated at 6 months to reflect favorable and unfavorable outcomes. The covariate of interest is a randomization assignment.

SECONDARY OUTCOMES:
Inpatient mortality | randomization to hospital discharge typically 2 weeks.
  We will assess the inpatient mortality of the participants. We will note the time from admission to death or discharge.
  The secondary outcome (inpatient mortality) will be analyzed using two approaches. The primary analysis model will be a logistic regression model where the outcome of interest is the vitality status (alive or dead) at discharge. The covariate of interest is a randomization assignment. The secondary analysis will be a time-to-death analysis comparing the survival curves between the two randomized groups using a log-rank test.

OTHER OUTCOMES:
To compare delayed interventions to treat Intracranial pressure (ICP). | randomization to hospital discharge, typically 2 weeks.
  Surgical or medical ICP-related therapeutic interventions. Events of acute kidney injury, cerebral edema, and in-patient mortality, will be captured.

CONTACTS AND LOCATIONS:
Overall Officials: Akshitkumar Mistry, MD, Principal Investigator — Assistant Professor Term
Locations (1):
- University of Louisville Hospital, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Undecided
Timeframe for sharing undecided at this early stage